CLINICAL TRIAL: NCT05877729
Title: iVY: Comprehensive, Tailored, Technology-based Intervention to Improve Virologic Suppression Among Youth and Young Adults Living With HIV
Brief Title: Intervention for Virologic Suppression in Youth
Acronym: iVY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); AIDS Healthcare Foundation (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-37017; R01MH131415 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HIV/AIDS; Young Adult; Mobile Health; Mental Health Issue; Substance Use
Keywords: Young Adults; Telehealth; Health Disparity; HIV; Mobile App
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (Active Comparator): The Standard of Care (SOC) arm will include the current care delivery model: regularly scheduled visits with a healthcare provider and lab testing every 3-6 months or more/less frequently depending on the individual's HIV health outcomes (e.g., VL suppression) . At each assessment, the investigators will review participant responses to examine acute need for referral for medical, psychological, or substance use services. In between assessments, researchers will also do monthly check-ins to improve retention and check contact information.
  Interventions: Other: Standard of Care
- Intervention Arm: Video-Counseling+app (Experimental): The video-counseling+app arm will receive 12 brief weekly counseling sessions (given over 16 weeks) with a social worker, along with access to the WYZ app to use based on their needs. After 16 weeks, participants receive another assessment and based on VL, those in the video-counseling+app arm will be categorized as intervention responders or non-responders (responder= virologically suppressed; non-responder= virologically unsuppressed. Responders in video-counseling+app arm will continue to use the app only. Non-responders in the intervention arm will continue with intensified video-counseling+app for 16 more weeks.
  Interventions: Behavioral: Video-counseling+app

INTERVENTIONS:
Other: Standard of Care — The SOC arm will include the current care delivery model: regularly scheduled visits with a healthcare provider and lab testing every 3-6 months or more/less frequently depending on the individual's HIV health outcomes (e.g., VL suppression). At each assessment, the investigators will review 149 SOC participant responses to examine acute need for referral for medical, psychological, or substance use services. In between assessments, the investigators will also do monthly check-ins to improve retention and check contact information.
  Other Names: SOC
  Arms: Standard of Care Arm
Behavioral: Video-counseling+app — The intervention tailors the telehealth counseling according to the individual's needs. Tailoring occurs based on the participant's baseline MH, SU, and HIV knowledge/outcomes and assessment responses inform the sessions on these topics. Participants choose from a list identified in the menu sessions: HIV care, MH, SU, lifestyle, health, social support, family of origin, romantic and sexual relationships, self-identity and disclosure, subsistence needs, education and vocation, and a "wildcard" session.
  WYZ contains 3 main features: My Health, My Team, and My Community. Tailoring is achieved based on the individual's needs at a given time (e.g., My Community may be used more if social isolation is a barrier).
  Other Names: iVY
  Arms: Intervention Arm: Video-Counseling+app

SUMMARY:
The goal of this randomized clinical trial is to test the effect of a technology-based intervention with an Adaptive Treatment Strategy (ATS) among youth living with HIV (YLWH) (18-29 years old). This piloted and protocolized intervention combines: (1) brief weekly sessions with a counselor via a video-chat platform (video-counseling) to discuss mental health (MH), substance use (SU), HIV care engagement, and other barriers to care; and (2) a mobile health application (app) to address barriers such as ART forgetfulness and social isolation. Individuals who are not virologically suppressed will be randomized to video-counseling+app or standard of care (SOC). Through this study, the investigators will be able to:

Aim 1: Test the efficacy of video-counseling+app vs SOC on virologic suppression in YLWH.The investigators will compare HIV virologic suppression of those randomized to the intervention vs control arms at 16 weeks via an RCT.

Aim 2: Assess the impact of video-counseling+app vs SOC on MH and SU in YLWH. The investigators will evaluate the MH and SU differences between the intervention vs control arms at 16 weeks via an RCT.

Aim 3: Explore an ATS to individualize the intervention by assigning the:

1. virologic "non-responders" in the intervention arm to intensified video-counseling+app for 16 more weeks,
2. virologic "responders" in the intervention arm to continue only app use for 16 more weeks.

Researchers will compare the characteristics of virologic responders and non-responders to the intervention, individualization of the intervention based on these variables, and linkage to MH and SU treatment services among those in need to see if delivery of care is enhanced and impact on virologic suppression.

DETAILED DESCRIPTION:
In the US, youth and young adults living with HIV (YLWH) have the lowest level of virologic suppression compared to older age groups and experience significant health disparities with regard to HIV treatment initiation and clinical outcomes. Additionally, mental health (MH) and substance use (SU) impact every step of the HIV care continuum from diagnosis to virologic suppression and exacerbate socioeconomic challenges of linkage and sustained access to healthcare.

The proposed study aims to address these barriers in a tailored manner using a differentiated care approach that is "youth-friendly". The iVY intervention is grounded in the Information Motivation Behavioral Skills (IMB) Model and developed with and for YLWH using a Human-Centered Design (HCD) approach. The goal is to test the effect of the technology-based intervention with differing levels of resource requirements (i.e., financial and personnel time) in a randomized clinical trial (RCT) with an Adaptive Treatment Strategy (ATS) among YLWH (18-29 years old). Using pre-defined algorithms, ATSs adapt a treatment to an individual's unique and changing needs as opposed to a one-size-fits-all approach.

Video-counseling will be delivered by clinical social workers trained to provide MH and SU counseling to YLWH. Video-counseling sessions will focus on the needs of the participant and potential linkage to further MH and SU treatment, as needed. The app will allow for medication management, identification of community resources, and online networking with other YLWH. Therefore, the primary goal of this approach is to address important, distinct, and changing barriers to HIV care engagement (e.g., MH, SU, forgetting, social isolation) among YLWH.

HIV virologic suppression (primary outcome) will be evaluated using home-collected Hemaspot test. To increase generalizability and geographic, demographic, and economic diversity and decrease logistics- or stigma-related barriers to research participation, all study activities will be conducted remotely. This study will provide valuable data about the characteristics of virologic responders and non-responders to the intervention, individualization of the intervention based on these variables, and linkage to MH and SU treatment services among those in need.

ELIGIBILITY:
Inclusion Criteria:

1. 18-29 years of age
2. HIV seropositive
3. Live and receive HIV care in California or Florida
4. Diagnosed with HIV more than 3 months ago
5. HIV VL test result of ≥20 copies at some point in the last 12 months (excluding tests within 3 mo of diagnosis)
6. Able to speak English
7. Have access to smartphone

Exclusion Criteria:

1. Unable or unwilling to provide consent.
2. Evidence of severe cognitive impairment, active psychosis, or substance use that may impede ability to provide informed consent during the consent process.
3. Those with a history of hemophilia or unable to conduct finger prick at home for the HIV viral load testing.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV Viral Load Suppression Comparison Evaluated Using Home-collected Hemaspot Device | 16 weeks
  Investigators will compare HIV virologic suppression of those randomized to the intervention vs control arm. HIV virologic suppression will be evaluated using home collected Hemaspot test.

SECONDARY OUTCOMES:
Clinical Impact: Frequency of Substance Use Comparison | 16 weeks
  Compare intervention and standard of care arms reported substance use at 16 weeks using Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), a 10-item question test administered through an online survey to measure frequency of participants' substance use. Higher score indicates high frequency of substance use.
Severity of Substance Use Comparison | 16 weeks
  Compare substance use scores in intervention and standard of care arms at 16 weeks using the Drug Abuse Screening Test (DAST), a 10-item questionnaire administered through an online survey to measure severity of participants' substance use. Responses are summed. Scoring (0-10);0-2 Low substance use, 9-10 Severe substance use. Higher score indicates higher severity of substance use.
Clinical Impact: Alcohol Use Comparison | 16 weeks
  Compare standard of care and intervention arms' alcohol use at 16 weeks using the Alcohol Use Disorder Test (AUDIT), a 10-item questionnaire administered through an online survey to measure severity of participants' alcohol use. Responses are summed. Scoring range is 0-20+; 0-7 Low alcohol use, 20+ High dependence. Higher score indicates higher alcohol misuse.
Clinical Impact: Depression Comparison | 16 weeks
  Compare intervention and control arms' depression scores at 16 weeks using the Patient Health Questionnaire (PHQ-9), a 9-item Likert scale score (0- 3) 0 "not at all", 3 "nearly every day". Responses are summed. Scores will have a range of 0-27. PHQ-9 scores of > 10 are associated with moderate to severe depression. Higher scores indicates more depressive symptoms.
Clinical Impact: PTSD (Post Traumatic Stress Disorder) Comparison | 16 weeks
  Compare intervention and standard of care arms self-reported PTSD symptom scores from baseline to 16 weeks using the Psychopathy Checklist-revised (PCL-5), a 20-item Likert questionnaire administered through an online survey. Scoring: 0 points for "not at all", 1 point for "a little bit", 2 points for "moderately", 3 points for "quite a bit", 4 points for "extremely". Scores will have a range of 0-80. Responses are summed. Higher score indicates more trauma.
Clinical Impact: Anxiety Comparison | 16 weeks
  Compare intervention and standard of care arms on self-reported anxiety scores measured at 16 weeks using Generalized Anxiety Disorder (GAD-7), a 7-item measure with scores from 0-21. A higher level score indicates more anxiety. Scores are summed and administered via online survey. Higher score indicates more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Parya Sabari, PharmD, Principal Investigator — UCSF School of Medicine, Division of Prevention Science
Locations (1):
- Division of Prevention Science, Center for AIDS Prevention Studies (CAPS), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saberi P, Ming K, Dawson-Rose C. What does it mean to be youth-friendly? Results from qualitative interviews with health care providers and clinic staff serving youth and young adults living with HIV. Adolesc Health Med Ther. 2018 Apr 24;9:65-75. doi: 10.2147/AHMT.S158759. eCollection 2018. PMID 29731672
- [Background] Wootton AR, Legnitto DA, Gruber VA, Dawson-Rose C, Neilands TB, Johnson MO, Saberi P. Telehealth and texting intervention to improve HIV care engagement, mental health and substance use outcomes in youth living with HIV: a pilot feasibility and acceptability study protocol. BMJ Open. 2019 Jul 16;9(7):e028522. doi: 10.1136/bmjopen-2018-028522. PMID 31315868
- [Background] McCuistian C, Wootton AR, Legnitto-Packard D, Gruber VA, Dawson-Rose C, Johnson MO, Saberi P. Addressing HIV care, mental health and substance use among youth and young adults in the Bay Area: description of an intervention to improve information, motivation and behavioural skills. BMJ Open. 2021 Apr 8;11(4):e042713. doi: 10.1136/bmjopen-2020-042713. PMID 38058024
- [Background] Saberi P, McCuistian C, Agnew E, Wootton AR, Legnitto Packard DA, Dawson-Rose C, Johnson MO, Gruber VA, Neilands TB. Video-Counseling Intervention to Address HIV Care Engagement, Mental Health, and Substance Use Challenges: A Pilot Randomized Clinical Trial for Youth and Young Adults Living with HIV. Telemed Rep. 2021 Jan 7;2(1):14-25. doi: 10.1089/tmr.2020.0014. eCollection 2021. PMID 33575683
- [Background] Erguera XA, Johnson MO, Neilands TB, Ruel T, Berrean B, Thomas S, Saberi P. WYZ: a pilot study protocol for designing and developing a mobile health application for engagement in HIV care and medication adherence in youth and young adults living with HIV. BMJ Open. 2019 May 5;9(5):e030473. doi: 10.1136/bmjopen-2019-030473. PMID 31061063
- [Background] Saberi P, Lisha NE, Erguera XA, Hudes ES, Johnson MO, Ruel T, Neilands TB. A Mobile Health App (WYZ) for Engagement in Care and Antiretroviral Therapy Adherence Among Youth and Young Adults Living With HIV: Single-Arm Pilot Intervention Study. JMIR Form Res. 2021 Aug 31;5(8):e26861. doi: 10.2196/26861. PMID 34463622
- [Derived] Saberi P, Stoner MCD, McCuistian CL, Balaban C, Ming K, Wagner D, Chakraborty B, Smith L, Sukhija-Cohen A, Neilands TB, Gruber VA, Johnson MO. iVY: protocol for a randomised clinical trial to test the effect of a technology-based intervention to improve virological suppression among young adults with HIV in the USA. BMJ Open. 2023 Oct 6;13(10):e077676. doi: 10.1136/bmjopen-2023-077676. PMID 37802624